CLINICAL TRIAL: NCT04052217
Title: Does Size Matter: A Single Case Experimental Design of Limiting the Depth of Penetration During Intercourse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: HR-16/17-2018
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Peyronie Disease
MeSH Terms: conditions — Penile Induration

STUDY DESIGN:
Intervention Model Description: Single Case Experimental Design
Who Masked: Participant
Masking Description: Masking of female participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Ring (Other): "Normal" intercourse with very thin (less than 0.5cm) ring randomised to either 3, 4 or 5 episodes of intercourse (Phase A)
  Interventions: Device: Penile Ring
- 1" RIng (Experimental): Intercourse wearing a 1" ring. Randomised to either 3, 4, or 5 episodes of intercourse (Phase B)
  Interventions: Device: Penile Ring
- 1.5" Ring (Experimental): Intercourse wearing a 1.5" ring randomised to either 3, 4, or 5 episodes of intercourse (Phase C)
  Interventions: Device: Penile Ring
- 2" Ring (Experimental): Intercourse with a 2" ring randomised to either 3, 4, or 5 episodes of intercourse (Phase D)
  Interventions: Device: Penile Ring

INTERVENTIONS:
Device: Penile Ring — Penile Ring at base of penis

SUMMARY:
Our hypothesis is that reducing the length of the penis does not lead to loss of sexual satisfaction or emotional closeness in the female partner. This will be investigated by a single case experimental design in 12 couples.

DETAILED DESCRIPTION:
The investigators will conduct a single case experimental design (SCED), in which a woman acts as her own control with a reversal design between randomly allocated phases. These include a control phase (A) and phases with various sizes of penile rings (B, C, and D).

The male participant will be asked to measure the length and girth of their erect penis using standardized instructions and flexible tape measure before the start of the experiment. This will partly determine the inner circumference of the ring provided. The male participant will be given instructions on how to use the penile rings and ensure that the female participant is blind to the size of the ring used.

There will be randomization (a) to the phase (the size of ring) and (b) the number of times of intercourse within a phase. The male partner will be blind to ratings made by the female partner. There is no carry over effect from one phase to another. The randomization of the phase means less guessing of the size of the ring, and less interaction with moderators (e.g. menstrual cycle, alcohol, holiday or life events randomly spread across phases). In a SCED, one then replicates in Case 2, Case 3 etc and a meta-analysis is conducted of all the single cases.

Randomisation will occur to either

1. Phase A "Normal" intercourse with very thin (less than 0.5cm) ring randomised to either 3, 4 or 5 episodes of intercourse)
2. Phase B - 1" ring randomised to either 3, 4, or 5 episodes of intercourse)
3. Phase C - 1.5" ring randomised to either 3, 4, or 5 episodes of intercourse)
4. Phase D - 2" ring randomised to either 3, 4, or 5 episodes of intercourse) The male partner will be kept informed by text or email or phone (whichever is convenient) of when to change the size of ring and the number of times it should be used. The female partner will be asked to be blind to the size of ring used after each episode of intercourse. Blindness will be tested by asking if the female partner "saw" the size of the ring or whether she was able to guess when a change in the size of the ring occurred.

Measures:

The investigators will use a Visual Analogue Scale (0-100) for the female participant ratings of (a) sexual pleasure and (b) how emotionally connected she felt to her partner (c) any adverse experiences.

The female participant will be asked to rate the degree of change (positive or negative) that would be significant for them e.g. a drop of rating 65 to 45) The female participant will be asked to rate satisfaction and emotional closeness as soon as possible after intercourse. The investigators will ask all participants to enter the data directly onto web based capture of data. This will be anonymized so that they will be identified by a character.

The male participant will be asked to confirm the size of the ring used and any other comments.

ELIGIBILITY:
Inclusion Criteria:

1. Heterosexual couples in a stable relationship (defined as 6 months or more)
2. Having regular intercourse (defined as on average twice a week).

Exclusion Criteria:

1. Any current sexual dysfunction in either partner
2. Any current emotional disorder in either partner
3. Men with a micro-penis

Min Age: 18 Years | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Overall Sexual Pleasure on a Visual Analogue Scale | Change between Control phase (A) and phase B, C, or D through study completion, on average 8 weeks
  Overall Sexual Pleasure on a Visual Analogue Scale between 0-100

SECONDARY OUTCOMES:
Sexual Pleasure from Intercourse on a Visual Analogue Scale | Change between Control phase (A) and phase B, C, or D through study completion, on average 8 weeks
  Sexual pleasure from intercourse alone on a Visual Analogue Scale between 0-100
Emotional Connection on a Visual Analogue Scale | Change between Control phase (A) and phase B, C, or D through study completion, on average 8 weeks
  Emotional Connection on a Visual Analogue Scale between 0-100

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Anxiety Disorders and Trauma, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All original data
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 10 years